CLINICAL TRIAL: NCT00004217
Title: A Phase II Study of Daunomycin and ARA-C Given by Continuous IV Infusion With PSC-833 for Previously Untreated Non-M3 Acute Myeloid Leukemia (AML) in Patients of Age 56 or Older
Brief Title: S9918 PSC 833, Daunorubicin, and Cytarabine in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S9918; S9918 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-01-28; First posted 2004-06-18 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Filgrastim; sargramostim; Cytarabine; Daunorubicin; valspodar

INTERVENTIONS:
Biological: filgrastim — 5 μg/kg/day IV or SC
Biological: sargramostim — 5 μg/kg/day IV or SC starting d 15
Drug: cytarabine — Ara-C continuous IV: Hours 2.5 - 170.5 before PSC-833
Drug: daunorubicin hydrochloride — continuous IV: Hours 2 - 74 before PSC-833
Drug: valspodar — 2 mg/kg load IV over 2 hrs (loading); 10 mg/kg/day Continuous hours 0 - 96

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. PSC 833 may help chemotherapy drugs kill more cancer cells by making them more sensitive to the drugs.

PURPOSE: Phase II trial to study the effectiveness of PSC 833, daunorubicin, and cytarabine in treating older patients who have newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of daunorubicin and cytarabine by continuous infusion and PSC 833 in patients over age 56 with newly diagnosed acute myeloid leukemia. II. Determine the frequency and severity of toxicities of this regimen in these patients. III. Determine the frequency and prognosis of functional and phenotypic P-glycoprotein expression, cytogenetics, and pharmacokinetics in this population.

OUTLINE: This is a multicenter study. Patients receive induction chemotherapy consisting of PSC 833 IV over 2 hours on day 1, then continuously for 96 hours; daunorubicin IV continuously on days 1-3; and cytarabine IV continuously on days 1-7. Filgrastim (G-CSF) or sargramostim (GM-CSF) is administered subcutaneously (SQ) or IV beginning on day 15 and continuing until blood counts recover or day 21. If patients do not achieve complete remission after one course, a second course is administered. Patients who achieve A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status after 1 or 2 courses of induction chemotherapy proceed to consolidation therapy, which begins upon recovery from induction therapy. Consolidation therapy consists of PSC 833 over 2 hours on day 1, daunorubicin IV over 1-5 minutes on days 1 and 2, and cytarabine IV continuously on days 1-5. Treatment repeats for a total of 2 courses. Patients are followed every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 20-55 patients will be accrued for this study within 8-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Morphologically confirmed acute myeloid leukemia (AML) No M3 AML or blastic phase chronic myelogenous leukemia Must be registered on protocols SWOG-9007 and SWOG-9910

PATIENT CHARACTERISTICS: Age: 56 and over Performance status: Zubrod 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT/SGPT no greater than 4 times ULN Renal: Creatinine no greater than 1.5 times ULN Creatinine clearance greater than 40 mL/min Cardiovascular: LVEF at least 50% by MUGA or echocardiogram No unstable cardiac arrhythmias or angina Other: Not pregnant or nursing Fertile patients must use effective contraception No other malignancy within the past 5 years except: Adequately treated basal cell or squamous cell skin cancer Carcinoma in situ of the cervix Adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for acute leukemia Prior hydroxyurea to control high cell counts allowed At least 30 days since prior low dose cytarabine (less than 100 mg/m2/day) for myelodysplastic syndrome and recovered Single dose of prior or concurrent (with induction chemotherapy) intrathecal chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2000-02; Primary Completion 2001-05 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
response | after induction therapy is completed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Chauncey, MD, PhD, Study Chair — VA Puget Sound Health Care System
Locations (90):
- United States (89):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844